CLINICAL TRIAL: NCT05679882
Title: Effects of Natural Sounds on Attention Restoration Outdoors
Acronym: NEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanyang Technological University (Other)
Collaborators: National Research Foundation, Singapore (Other Government); Ministry of National Development, Singapore (Other Government); Housing and Development Board, Singapore (Other Government)
Responsible Party: Principal Investigator, Georgios CHRISTOPOULOS, Associate Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COT-V4-2020-1-S004
Record Dates: First submitted 2022-09-05; First posted 2023-01-11 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Cognitive Fatigue; Mental Fatigue; Behavioral Performance; Heart Rate Variability; Positive and Negative Affect; Inhibition, Psychological; Working Memory; Perceived Restoration
MeSH Terms: conditions — Mental Fatigue; Inhibition, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outdoor Environment (Active Comparator): Exposure to outdoor environmental noise
  Interventions: Other: No Masking Sounds
- Outdoor Environment with Machine-Learning Selected Masking Sounds (Experimental): Exposure to outdoor environmental noise and masking sounds
  Interventions: Other: Masking Sounds

INTERVENTIONS:
Other: Masking Sounds — Masking sounds will be played from outdoor speakers.
  Arms: Outdoor Environment with Machine-Learning Selected Masking Sounds
Other: No Masking Sounds — No masking sounds will be played from outdoor speakers.
  Arms: Outdoor Environment

SUMMARY:
This study aims to examine whether listening to natural sounds in a noisy outdoor environment compared to no natural sounds influences behavioural, cognitive, affective, and physiological markers.

DETAILED DESCRIPTION:
The investigators hypothesize that listening to natural sounds has restorative effects on attention by supporting greater use of involuntary attention. This generates the prediction that exposure to natural sounds in the context of a noisy outdoor environment will have greater restorative effects on attention (i.e., physiological, affective, cognitive, and behavioural) as compared to the control group (exposed to environmental noise only). Individual differences (i.e., age, gender, caffeine and food intake, body mass index, skin temperature, noise sensitivity, sleep quality, baseline physiology and behavioural performance) will be examined and accounted for. Environmental factors (i.e., outdoor humidity, temperature, and noise) will also be accounted for.

ELIGIBILITY:
Inclusion Criteria:

* Singapore-based
* Non-clinical
* 18-35years

Exclusion Criteria:

* Individuals with hearing difficulties or failing to meet the minimal threshold for normal hearing
* Individuals with a history of ear, developmental, neurological, or psychiatric disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Reverse Corsi Task (Change) | baseline and up to 60 mins after sound intervention
  Change in Span and Reaction Time
Go/NoGo Task (Change) | baseline and up to 60 mins after sound intervention
  Change in Accuracy and Reaction Time
Change in Heart Rate Variability | 1 day (during fatiguing task and sound intervention)
  Electrocardiograph and photoplethysmograph (Change)
Positive and Negative Affect Schedule - Expanded Form | up to 60 mins after sound intervention
  Positive and Negative Affect Score
Fatigue State Questionnaire (Change) | baseline and up to 60 mins after sound intervention
  Change in Fatigue State Questionnaire Score

SECONDARY OUTCOMES:
Perceived Restorativeness Soundscape Scale | up to 60 mins after sound intervention
  Perceived Restorativeness Soundscape Scale Score

CONTACTS AND LOCATIONS:
Locations (1):
- Cultural Science Innovations, Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No